CLINICAL TRIAL: NCT03965169
Title: Incidence and Risk Factors of Postoperative Pressure Injury in Patients Undergoing Prone Spinal Surgery
Brief Title: Postoperative Pressure Injury in Patients Undergoing Prone Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pressure injury
Record Dates: First submitted 2019-04-25; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-04

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing prone spinal surgery (Experimental): Patients undergoing elective spinal surgery in prone position under general anesthesia, which is performed by neurosurgeons in Seoul National University Hospital
  Interventions: Procedure: Prone spinal surgery

INTERVENTIONS:
Procedure: Prone spinal surgery — spinal surgery in prone position under general anesthesia

SUMMARY:
Patients undergoing surgery under general anesthesia are susceptible to pressure-induced soft tissue damage because there is no change in posture over an extended period of time. In particular, when the patient is in a prone position, unlike the supine position, the bony protruding portion of the front side must support the weight, which is more vulnerable to pressure injury. Previous studies have shown that the incidence of pressure injury during surgery varied from 5% to 66% and was more likely to occur in patients with long operating times, prone position, obesity, and poor skin condition. These pressure injuries increase postoperative complications, length of stay, and medical costs. Therefore, the investigators analyze the incidence of pressure injury in prone position and re-examine the risk factors of pressure injury.

DETAILED DESCRIPTION:
All of the anesthetic and surgical procedures performed on the subject during the period from the time the subject enters the operating room to the time the subject go to the recovery room are the same as those for the existing spine surgery. Immediately after entering the operating room, immediately before going to the recovery room, and at postoperative day 1 and 2, the patient's systemic skin condition is assessed to determine whether pressure damage has occurred. The primary endpoint is the incidence of pressure injury in the subject compared with the incidence of pressure injury in previous studies. To identify the risk factors for the occurrence of pressure injury, the investigators will statistically analyze the data collected with the assumption that this is related.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing elective spine surgery in prone position under general anesthesia

Exclusion Criteria:

* Pre-existence of pressure injury

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pressure injury | From end of surgery to postoperative day 2
  The pressure injury after prone spine surgery will be identified and evaluated using "Pressure injury staging illustration - National Pressure Ulcer Advisory Panel" at end of surgery, postoperative day 1 and 2. The prevalence of pressure injury will be calculated by dividing the number of patients with pressure injury by the total number of patients.

SECONDARY OUTCOMES:
Site of pressure injury | From end of surgery to postoperative day 2
  The pressure injury after prone spine surgery will be identified and evaluated using "Pressure injury staging illustration - National Pressure Ulcer Advisory Panel" at end of surgery, postoperative day 1 and 2. The site of pressure injury will be categorized as head, chest, abdomen, arm, leg and others.
Grade of pressure injury | From end of surgery to postoperative day 2
  he pressure injury after prone spine surgery will be identified and evaluated using "Pressure injury staging illustration - National Pressure Ulcer Advisory Panel" at end of surgery, postoperative day 1 and 2. The grade of pressure injury will be categorized as 1, 2, 3, and 4 according to the definition in "Pressure injury staging illustration - National Pressure Ulcer Advisory Panel".

CONTACTS AND LOCATIONS:
Overall Officials: Hyongmin Oh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin S, Hey HWD, Lau ETC, Tan KA, Thambiah JS, Lau LL, Kumar N, Liu KG, Wong HK. Prevalence and Predictors of Pressure Injuries From Spine Surgery in the Prone Position: Do Body Morphological Changes During Deformity Correction Increase the Risks? Spine (Phila Pa 1976). 2017 Nov 15;42(22):1730-1736. doi: 10.1097/BRS.0000000000002177. PMID 28368987
- [Background] Schoonhoven L, Defloor T, Grypdonck MH. Incidence of pressure ulcers due to surgery. J Clin Nurs. 2002 Jul;11(4):479-87. doi: 10.1046/j.1365-2702.2002.00621.x. PMID 12100644
- [Background] Kim JM, Lee H, Ha T, Na S. Perioperative factors associated with pressure ulcer development after major surgery. Korean J Anesthesiol. 2018 Feb;71(1):48-56. doi: 10.4097/kjae.2018.71.1.48. Epub 2017 Jul 4. PMID 29441175
- [Background] Scarlatti KC, Michel JL, Gamba MA, de Gutierrez MG. [Pressure ulcers in surgery patients: incidence and associated factors]. Rev Esc Enferm USP. 2011 Dec;45(6):1372-9. doi: 10.1590/s0080-62342011000600014. Portuguese. PMID 22241195